CLINICAL TRIAL: NCT00978588
Title: Comparison of 6% Hydroxyethyl Starch 130/0.4 With 5% Albumin as Priming Solution for Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2007-0429
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Mitral Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Hydroxyethyl Starch Derivatives; Albumins

ARMS (2):
- HES 130/0.4 (Experimental)
  Interventions: Drug: 6% hydroxyethyl starch 130/0.4 and 5% albumin
- 5% albumin (Active Comparator)
  Interventions: Drug: 6% hydroxyethyl starch 130/0.4 and 5% albumin

INTERVENTIONS:
Drug: 6% hydroxyethyl starch 130/0.4 and 5% albumin — Injection of 6% hydroxyethyl starch 130/0.4 and 5% albumin as priming solution for cardiopulmonary bypass

SUMMARY:
Comparison of 6% hydroxyethyl starch 130/0.4 with 5% albumin as priming solution for cardiopulmonary bypass

ELIGIBILITY:
Inclusion Criteria:

* Mitral valvular heart disease

Exclusion Criteria:

* Status of Infection
* Re-operation
* Liver failure
* Renal disease
* Administration of steroid

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
the pure effect of priming solutions | after CPB

CONTACTS AND LOCATIONS:
Overall Officials: Young Lan Kwak, M.D.,PhD,, Principal Investigator — Severance Hospital